CLINICAL TRIAL: NCT00224354
Title: Treatment of Chronic Lymphocytic B-Leukemia (B-CLL) With Human IL-2 Gene Modified and Human CD40 Ligand-Expressing Autologous Tumor Cells After Depletion of Regulatory T Cells
Brief Title: Lymphocytic B-Leukemia (B-CLL) w/Human IL-2 Gene Modified & Human CD40 Ligand-Expressing Autologous Tumor Cells
Acronym: CLONTAK
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, George Carrum, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17656; CLONTAK
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: CHRONIC LYMPHOCYTIC B-LEUKEMIA
Keywords: LYMPHOCYTIC; B-LEUKEMIA; B-CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Interleukin-2; CD40 Ligand; denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: IL-2 secreting and hCL4OL-expressing autologous B-CLL cells — Patients will be treated with six subcutaneous injections of their IL-2-secreting and hCD40L-expressing autologous B-CLL cells, separated by one to two weeks in an immunological treatment window
Biological: IL-2 — subcutaneous (SC) injections of autologous leukemic cells modified ex vivo to secrete human interleukin-2 (hIL-2) and to express human CD40 ligand (hCD40L).
Biological: CD40L — subcutaneous (SC) injections of autologous leukemic cells modified ex vivo to secrete human interleukin-2 (hIL-2) and to express human CD40 ligand (hCD40L).
Drug: ONTAK — an interleukin-2 immunotoxin directed to the CD25 antigen (denileukin diftitox, ONTAK
Biological: immunotoxin dose — Days 0, 2, and 4 (18 ug/kg) i.v
  Other Names: ONTAK

SUMMARY:
In the laboratory, we will put a special gene into cancer cells that have been taken from the subject. This gene will make the cells produce interleukin 2 (IL-2), which may help the patient's immune system kill cancer cells. Also, we will use CD40 ligand (CD40L) with the IL-2. Studies of cancers in animals and in cancer cells that are grown in laboratories have suggested adding the CD40L helps the IL-2 work better. Some of these new cells will then be given back to the subject as a vaccine shot.

We believe that a part of the subject's immune system (cells called T-reg cells) might try to kill off these special cells. If the T-reg cells do that, the vaccine would not work as well or last as long. To try to avoid this, before the special cells are put back into the subject's body, we will give them an intravenous (IV) dose of IL-2 immunotoxin (called denileuk diftitox or ONTAK). ONTAK should get rid of some of the T-reg cells in the subject's body which should help the special cells work better and longer.

The purpose of this study is to learn the safety and cancer-fighting effects of using IL-2 with the vaccine.

DETAILED DESCRIPTION:
This is a phase I trial to assess the safety of depleting regulatory T (Treg) cells using 1-3 doses of an interleukin-2 immunotoxin directed to the CD25 antigen (denileukin diftitox, ONTAK) in chronic lymphocytic leukemia (B-CLL) patients, followed by six subcutaneous (SC) injections of autologous leukemic cells modified ex vivo to secrete human interleukin-2 (hIL-2) and to express human CD40 ligand (hCD40L). Patients will receive a fixed dose (2 x 10e7) of IL-2 secreting B-cells together with 2 x 10e7 hCD40L expressing B-cells, representing a safe, well tolerated and immunogenic dose in our previous dose escalation study.

All eligible patients will be treated with six injections. Any patient whose disease regresses after the administration of 6 injections may be offered further injections of tumor vaccine if sufficient vaccine is available. There will be no use of placebo or control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Pre Inclusion Eligibility Criteria: Proof of B-CLL diagnosis not in Richter's transformation

Eligibility Criteria:

* Manipulated B-CLL cells available (at least 6 injections)
* B-CLL with measurable disease, not in Richter's transformation
* Life expectancy greater than or equal to 10 weeks
* ECOG 0-2 (see Section 4.3 of the full protocol for details)
* Recovered from the toxic effects of all prior chemotherapy
* Absolute neutrophil count (ANC) greater than or equal to 500/mL
* Absolute lymphocyte count (ALC) greater than or equal to 200/mL
* Hemoglobin greater than or equal to 8 g/dL
* Platelet count greater than or equal to 50,000/mL
* Total bilirubin less than or equal to 1.5mg/dL -SGOT less than or equal to 2 x Normal
* Normal PTT -Creatinine less than 3 x Normal (age-related) or Creatinine clearance > 80mg/min/1.73m2
* Serum albumin level greater than or equal to 3 g/dl
* Must not have received treatment with other investigational agents within the last 4 weeks
* Practicing appropriate birth control during the study and for 3 months after the study is concluded.

Exclusion Criteria:

* Congestive heart failure
* Significant arrythmia or history of myocardial infarction
* Active CNS disease or a history of seizure
* Active infection / receiving antibiotics (other than prophylactic trimethoprim sulfamethoxazole
* Seropositive for HIV
* Pregnancy or lactation / will not use birth control methods
* Autoimmune disease (GvHD, immune thrombocytopenia-ITP or autoimmune hemolytic anemia-AIHA)
* Receiving immunosuppressive drugs
* Hypersensitivity to denileukin diftitox or any of its components: diphteria toxin, interleukin-2, or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety of (Treg) cells using interleukin-2 immunotoxin directed to the CD25 antigen in(B-CLL) patients, then six (SC) injections of autologous leukemic cells modified to secrete (hIL-2) and to express (hCD40L). | 15 years
To obtain preliminary data on the anti-tumor effects of this treatment regimen. | 15 years

SECONDARY OUTCOMES:
determine whether MHC-restricted or unrestricted anti-tumor immune responses are induced and sustained by the combination of Treg cell depletion and SC injections of B-CLL cells, which have been modified ex vivo to secrete hIL-2 and to express hCD40L | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: GEORGE CARRUM, MD, Principal Investigator — Baylor College of Medicine; Malcolm K Brenner, MD, Study Director — Baylor College of Medicine